CLINICAL TRIAL: NCT05503927
Title: Wegovy® (Semaglutide 2.4 mg) Database Study: A Population-based Cohort Study to Investigate Safety Outcomes of Exposure to Wegovy During Pregnancy
Brief Title: A Study to Evaluate the Safety of Exposure to Wegovy During Pregnancy
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-4971; U1111-1273-4411 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-08-10; First posted 2022-08-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants Exposed to Wegovy: Pregnant participants exposed to Wegovy during the first trimester (T1) (that is, estimated conception date - 35 days through <14 weeks gestational age [WGA]) and their linked infants will be observed in this retrospective observational study.
  Interventions: Other: No Intervention
- Participants Exposed to Anti-obesity Medication (AOM): Pregnant participants exposed to other Anti-obesity Medication (AOM) (phentermine, diethylpropion, benzphetamine, phendimetrazine, orlistat, or bupropion/naltrexone) during the first trimester (start of exposure identification window based on five times the half-life of each AOM through <14 WGA) and their linked infants will be observed in this retrospective observational study.
  Interventions: Other: No Intervention
- Overweight/Obese Participants: Pregnant participants with obesity or overweight and 1 or more comorbid condition without exposure to Wegovy or other AOM during pregnancy will be observed in this retrospective observational study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study, therefore no intervention is used.

SUMMARY:
This is an observational, retrospective, cohort study using administrative insurance claims data. The aim of this non-interventional study (NIS) is to compare maternal, fetal and infant outcomes of women exposed to Wegovy during pregnancy to a reference population not exposed to Wegovy, so that participants and healthcare providers can make informed treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a pregnancy end event on a medical claim (example, live birth, stillbirth, or spontaneous abortion) during the pregnancy identification period (that is, 04 June 2021 - 17 February 2027).
* Aged 15-45 and female on the date of the last menstrual period (LMP).
* Continuous enrolment in the database with medical and pharmacy benefits for at least 6 months prior to the date of LMP through 42 days after the pregnancy end date.
* Among the pregnancies that meet the inclusion criteria, three main cohorts of interest and two sub cohorts will be identified (one Wegovy-exposed cohort and two comparison cohorts):
* Wegovy-exposed- for greater than or equal to 1 day of Wegovy exposure from estimated conception date (LMP +14) - 35 days to end of pregnancy.
* Other AOM-exposed- greater than or equal to1 day of phentermine, diethylpropion, benzphetamine, phendimetrazine, orlistat, or bupropion/naltrexone exposure, defined as the following:
* Benzphetamine, diethylpropion, orlistat, or phendimetrazine exposure from estimated conception date-1 day to end of pregnancy.
* Phentermine or bupropion/naltrexone exposure from estimated conception date- 5 days to end of pregnancy.
* Cohort with Overweight/Obesity-
* Greater than or equal to 1 diagnosis code for obesity or BMI greater than or equal to 30 kilogram per meter square (kg/m^2) on a medical claim during the six month pre-pregnancy period.
* Greater than or equal to 1 diagnosis code for BMI greater than or equal to 27 kg/m^2 or less than 30 kg/m^2 on a medical claim and greater than or equal to 1 non-diagnostic medical claim for dyslipidemia, type 2 diabetes mellitus, or hypertension during the six month pre-pregnancy period.
* No exposure to Wegovy or other AOM during the defined exposure window in pregnancy.
* Among Wegovy-exposed and Other AOM-exposed pregnancies, the subset with first trimester exposures will be identified as those with greater than or equal to 1 days of exposure at < less than 14 WGA.

Exclusion Criteria:

* Pregnancies exposed to other glucagon-like peptide-1 receptor agonist (GLP-1 RA) during the exposure identification window (estimated conception date - 35 days through pregnancy end date).
* Pregnancies with exposure to both Wegovy and other AOM during the exposure identification window (estimated conception date - 35 days through pregnancy end date).
* Pregnancies resulting in multiple infants will be excluded from the analysis of infant outcomes.

Ages: 15 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — This is a study of prenatal exposure to Wegovy in pregnant women.
Study Population: Pregnant participants exposed to Wegovy, other AOM and pregnant participants with obesity and overweight were observed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 1139 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Number of Infants with Major Congenital Malformation (MCM) | Birth up to 1 year of age
  Number of infants with MCM is defined as an abnormality of body structure or function that is present at birth, is of prenatal origin (that is, birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention.

SECONDARY OUTCOMES:
Number of Infants Experiencing Small for Gestational Age (SGA) Birth | Birth up to 1 year of age
  Number of infants experiencing small for gestational age is defined as weight at birth in less than (<) 10th percentile for sex and gestational age using standard growth charts for full and preterm live born infants.
Number of infants with Developmental Delay | Birth up to 1 year of age
  Infant development delay will be defined as infants with evidence of one or more of the following outcomes in the first year of life: delayed milestone in childhood, other lack of normal physiological development, special screening for developmental disabilities.
Number of Infants With Postnatal Growth Deficiency | Birth up to 1 year of age
  Number of infants with adverse postnatal growth will be defined as infants with evidence of the following outcomes in the first year of life: abnormal weight gain (insufficient or excessive weight gain), short stature, failure to thrive.
Number of Pregnant Participants Experiencing Stillbirth | up to 37 weeks of gestational age
  Number of pregnant participants experiencing still birth is defined as an involuntary fetal loss occurring at greater than or equal to (>=20) WGA.
Number of Pregnant Participants Experiencing Spontaneous Abortion (SAB) | up to 37 weeks of gestational age
  Number of pregnant participants experiencing SAB is defined as an involuntary fetal loss or the expulsion of the products of conception occurring at <20 WGA.
Number of Pregnant Participants With Preterm Delivery | Up to 37 weeks of gestational age
  Preterm birth is defined as a live birth occurring at <37 WGA.
Number of Pregnant Participants With Pre-eclampsia/eclampsia | Up to 37 weeks of gestational age
  Pre-eclampsia/eclampsia is defined as new onset of hypertension with proteinuria occurring at >=20WGA through the six weeks following pregnancy end.

CONTACTS AND LOCATIONS:
Overall Officials: (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com